CLINICAL TRIAL: NCT07278531
Title: Adaptive Dietary Intervention (ADI) Leveraging Continuous Glucose Monitoring for Asian Americans With Type 2 Diabetes
Brief Title: Adaptive Dietary Intervention (ADI) for Asian Americans With Type 2 Diabetes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-01868
Record Dates: First submitted 2025-12-03; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- CGM Alone (Experimental): CGM only for weeks 1-4, continue with CGM only for weeks 4-12; this arm includes individuals who achieved the glycemic control goal at week 4.
  Interventions: Device: Continuous Glucose Monitoring (CGM)
- CGM Alone, then CGM-GEM (Experimental): CGM only for weeks 1-4; then CGM augmented with CEM for weeks 4-12; this arm includes individuals who did NOT achieve the glycemic control goal at week 4.
  Interventions: Device: Continuous Glucose Monitoring (CGM); Behavioral: Adaptive dietary intervention (GEM)
- Standard of Care (SC) (No Intervention): Usual diabetes care. Current standard of care will be followed, including regular appointments (2-4 times/year) with A1c monitoring, medication titration, and screening for diabetes complications.

INTERVENTIONS:
Device: Continuous Glucose Monitoring (CGM) — Participants will receive a walk-through for CGM use with the research staff, including insertion and initiation of CGM, alarm parameter settings, data sharing via LibreView, checking and reviewing CGM glucose values and trends via Libre app or CGM reader, and the relationship between food intake and CGM results.
  Arms: CGM Alone; CGM Alone, then CGM-GEM
Behavioral: Adaptive dietary intervention (GEM) — Adapted glycemic excursion minimization (CGM-GEM).
  Arms: CGM Alone, then CGM-GEM

SUMMARY:
The investigators will examine the feasibility, acceptability, and effect of an adaptive dietary intervention over 24 weeks (12-week intervention, 12-week follow-up) among Asian Americans with Type 2 diabetes. Participants (N=120; 60 Chinese Americans and 60 Vietnamese Americans) will be 2:1 randomized to one of two arms: adaptive dietary intervention or standard of care (SC). The intervention will begin with continued glucose monitoring (CGM) use only during weeks 0-4. At week 4, participants who achieve the glycemic control goal (at least an 8% increase in time in range [TIR] from baseline) will continue with the CGM alone during weeks 4-12 ("CGM Alone"); otherwise, culturally and linguistically adapted glucose excursion minimization (GEM) will be augmented with CGM ("CGM-GEM").

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants (N=120; 60 Chinese Americans and 60 Vietnamese Americans)
* Community-dwelling adults aged ≥ 18 with independent living;
* Diagnosed with T2D;
* Hb1Ac>7.0%
* Self-identified as first- or second-generation Chinese or Vietnamese immigrants;
* Able to communicate in English, Chinese, or Vietnamese. We will focus on Mandarin-, Cantonese- or English-speaking Chinese Americans because the two best-known and most-spoken variants of Chinese are Mandarin and Cantonese, who use the same writing system;
* Have a smartphone, iPad, tablet, or Apple watch

Exclusion Criteria:

* Taking hypoglycemia agents (e.g., insulin and sulfonylureas) with the major side effect of hypoglycemia that need close monitoring the occurrence of hypoglycemia to adjust/reduce medications to avoid future hypoglycemia.
* Taking medications that impede weight loss (e.g., prednisone) within the last 3 months.
* Currently pregnant, breastfeeding, or contemplating pregnancy within the next 6 months.
* Have serious physical complications (e.g., severe neuropathy cardiovascular disease, COPD/emphysema, osteoarthritis, or stroke) or mental disease (e.g., schizophrenia, bipolar disorder, manic depressive illness, severe depression, or active substance abuse).
* Have conditions that restrict diet, such as severe gastroparesis, ulcers, or food allergies. These conditions may need special dietary intervention.
* Undergoing treatment for cancer, as cancer treatment may impact the outcome of glucose changes.
* Have marked renal impairment (eGRF<45; CKD-3b), as renal impairment may needs special dietary intervention and they also may impact glucose changes.
* Are taking psychotropic medications that raise blood glucose (e.g., atypical antipsychotics).
* Are prior or current CGM users including both Dexcom and FreeStyle Libre and plan to continuously use these CGMs in the next 6 months.
* Are participating in another T2D intervention study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment Rate | Baseline
  Proportion of eligible participants who enroll in the trial.
Retention Rate | Week 24
  Proportion of recruited participants who complete the trial.
Glycated Hemoglobin (A1c) Level - Baseline | Baseline
Glycated Hemoglobin (A1c) Level - Week 12 | Week 12
Glycated Hemoglobin (A1c) Level - Week 24 | Week 24
Time in Range (TIR) - Baseline | Baseline
  "Time in range" (TIR) refers to the percentage of time a participant spends with their blood glucose levels within the target range.
Time in Range (TIR) - Week 12 | Week 12
  "Time in range" (TIR) refers to the percentage of time a participant spends with their blood glucose levels within the target range.
Time in Range (TIR) - Week 24 | Week 24
  "Time in range" (TIR) refers to the percentage of time a participant spends with their blood glucose levels within the target range.

CONTACTS AND LOCATIONS:
Overall Officials: Yaguang Zheng, PhD, RN, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 3 months to 5 years after publication, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: Yaguang.Zheng@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements. The informed consent form, clinical study report and analytic code will also be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Yaguang.Zheng@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.